CLINICAL TRIAL: NCT03557801
Title: Assessing the Impact of a Community Health Worker on Hispanic Women's Reported Measures of Processes of Care in the Screening Mammography Setting
Brief Title: Promotora Navigator - Culturally Appropriate Patient Navigator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lucy Spalluto, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 180276
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Results first posted 2019-07-31 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Screening Mammography; Community Health Worker
MeSH Terms: conditions — Breast Neoplasms | interventions — Community Health Workers; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care Mammography (Active Comparator): Immediately following consent and completion of the baseline assessment, women in the control arm will receive standard of care well woman screening. The control arm will receive screening results per standard of care protocol.
  Interventions: Other: Standard of Care Mammography
- Mammography with Community Health Worker (individual) (Experimental): Immediately following consent and completion of the baseline assessment, women in the intervention arm 1 will participate in a 20-30 minute educational session alone with the community health worker. Well woman screening will follow the educational session. The community health worker will be available to assist with questions and language interpretation as necessary. After standard delivery of screening results, the community health worker will contact these participants to answer any questions about their screening results and to assist with scheduling any additional tests necessary.
  Interventions: Behavioral: Mammography with Community Health Worker (individual)
- Mammography with Community Health Worker (group) (Experimental): Immediately following consent and completion of the baseline assessment, women in the intervention arm will participate in a 20-30 minute group educational session from the community health worker. Well woman screening will follow the educational session. The community health worker will be available to assist with questions and language interpretation as necessary. After standard delivery of screening results, the community health worker will contact these participants to answer any questions about their screening results and to assist with scheduling any additional tests necessary.
  Interventions: Behavioral: Mammography with Community Health Worker (group)

INTERVENTIONS:
Behavioral: Mammography with Community Health Worker (individual) — Immediately following consent and completion of the baseline assessment, alone with the community health worker. Well woman screening will follow the educational session. The community health worker will be available to assist with questions and language interpretation as necessary. After standard delivery of screening results, the community health worker will contact these participants to answer any questions about their screening results and to assist with scheduling any additional tests necessary.
  Arms: Mammography with Community Health Worker (individual)
Behavioral: Mammography with Community Health Worker (group) — Immediately following consent and completion of the baseline assessment, women in the intervention arm will participate in a 20-30 minute group educational session from the community health worker. Well woman screening will follow the educational session. The community health worker will be available to assist with questions and language interpretation as necessary. After standard delivery of screening results, the community health worker will contact these participants to answer any questions about their screening results and to assist with scheduling any additional tests necessary.
  Arms: Mammography with Community Health Worker (group)
Other: Standard of Care Mammography — Immediately following consent and completion of the baseline assessment, women in the control arm will receive standard of care well woman screening. The control arm will receive screening results per standard protocol.
  Arms: Standard of Care Mammography

SUMMARY:
Although there has been interval improvement in reducing disparity in mammography utilization in medically underserved communities since the 1990s, significant disparities persist and should be addressed. In the 40-65 year old age range, there is significant disparity in screening mammography utilization in Hispanic women compared to their white counterparts.

Culturally adapted patient-targeted healthcare interventions can help reduce ethnic inequalities in access to cancer screening programs. Promotoras, culturally appropriate patient navigators for the Hispanic community, have been shown to increase screening mammography rates in the Hispanic/Latino population.

However, there is little research exploring the interaction between these lay community health workers and community members. This proposal aims to assess this interaction by measuring the impact of a Promotora working with community members in either a group setting or individual setting. Understanding this interaction can lead to more effectively designed future community interventions. Primary outcomes in this study will include women's reported measures of interpersonal processes of care (communication and interpersonal style) during screening mammography care, trust in the healthcare system, and satisfaction with cancer screening care when compared to those receiving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Identifying as Hispanic ethnicity
* Age 40-64
* Tennessee resident

Exclusion Criteria:

* Personal history of breast cancer
* Current breast symptoms (palpable mass)

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Spalluto, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Matthew Walker Comprehensive Health Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Mammography With Community Health Worker (Group): Immediately following consent and completion of the baseline assessment, women in the intervention arm 2 will participate in a 20-30 minute group educational session from the community health worker. Well woman screening will follow the educational session. The community health worker will be available to assist with questions and language interpretation as necessary. After standard delivery of screening results, the community health worker will contact these participants to answer any questions about their screening results and to assist with scheduling any additional tests necessary.
Period: Overall Study
Arm/Group | Standard of Care Mammography | Mammography With Community Health Worker (Individual) | Mammography With Community Health Worker (Group)
Started | 34 | 33 | 33
Completed | 32 | 32 | 30
Not Completed | 2 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Mammography | Mammography With Community Health Worker (Individual) | Mammography With Community Health Worker (Group) | Total
Number analyzed (Participants) | 34 | 33 | 33 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (6.8) | 48.2 (7.3) | 47.3 (5.6) | 47.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 33 | 100
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 33 | 33 | 100
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Measures From Interpersonal Processes of Care Survey
Description: Selected scales (communication and interpersonal style) of the Interpersonal Processes of Care Survey will be the primary outcome. A total of 18 (corrected from orginal submission) questions will be administered. The questions are scored on a scale from 1-5 with higher scores indicating higher frequencies of the construct. The compiled scores will range from 5-90. Scales with negative associations (discrimination, hurried communication) will be reversed. Thus, higher scores for all items will indicate a more positive experience.
Time Frame: Approximately 2 weeks after consent/screening mammogram.
Population: Participants that completed the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care Mammography | Mammography With Community Health Worker (Individual) | Mammography With Community Health Worker (Group)
Number analyzed (Participants) | 32 | 32 | 30
score on a scale | 73 [70.5 to 79] | 78 [75 to 84] | 77 [72 to 85]

2. Secondary Outcome: Patient Reported Measures From the Distrust in the Healthcare System Scale. Reported at Baseline and Post Intervention. Also Reported as the Change Between Baseline and Intervention.
Description: Distrust will be measured with the Revised Healthcare System Distrust Scale. This 9 question scale is divided into two subscales: competence and values. The questions are scored on a scale from 1-5. The total score will range 5-45, with higher scores indicating higher levels of trust. Baseline distrust measured at time of initial consent/screening. Post-intervention distrust measured at time of post-survey which took place approximately 2 weeks after screening (varied as to when patient could be reached for survey). Difference in distrust is subtracts the baseline score from the post score.
Time Frame: Baseline, approximately 2 weeks after consent/screening mammogram.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Mammography | Mammography With Community Health Worker (Individual) | Mammography With Community Health Worker (Group)
Number analyzed (Participants) | 32 | 32 | 30
score on a scale
  Pre intervention | 32.5 (5.6) | 32.5 (4.9) | 33.6 (5.5)
  Post Intervention | 32.7 (4.5) | 33.7 (4.6) | 33.6 (4.6)

3. Secondary Outcome: Patient Reported Measures From the Satisfaction With Cancer Related Care Scale.
Description: Satisfaction with care will be measured with the Patient Satisfaction with Cancer-Related Care (PSCC) Measure. This is an 18 question measure. The questions are scored on a scale from 1-5. The total score will range 5-90, higher scores indicate higher satisfaction with care.
Time Frame: Approximately 2 weeks after consent/screening mammogram.
Population: Participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Mammography | Mammography With Community Health Worker (Individual) | Mammography With Community Health Worker (Group)
Number analyzed (Participants) | 32 | 32 | 30
score on a scale | 74.9 (6.6) | 78.1 (8.6) | 78.8 (5.3)

ADVERSE EVENTS:
Time Frame: 1 month.
Arm/Group | Standard of Care Mammography | Mammography With Community Health Worker (Individual) | Mammography With Community Health Worker (Group)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT03557801/Prot_SAP_000.pdf